CLINICAL TRIAL: NCT00448838
Title: Pilot Study of Gemcitabine, Oxaliplatin, and Cetuximab for Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Cetuximab, Gemcitabine, and Oxaliplatin in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20057548; SCCC-2005141 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20052717 (Other: Western Insitutional Review Board)
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Cetuximab — Cetuximab: an initial loading dose of 400 mg/m2 will be given followed by 250 mg/m2 administered weekly. Cetuximab will be given first followed by gemcitabine on the weeks the patient receives cytotoxic chemotherapy on day 1. Cetuximab will be given as a single agent on Day 8. The treatment will be given on two-week cycles.
  Other Names: C-225
Drug: Gemcitabine Hydrochloride — Gemcitabine 1000 mg/m2 IV day 1. The treatment will be given on two-week cycles.
  Other Names: Gemcitabine HCl
Drug: Oxaliplatin — Oxaliplatin 100 mg/m2 IV day 2. The treatment will be given on two-week cycles.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of pancreatic cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as gemcitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving cetuximab together with combination chemotherapy may kill more tumor cells.

PURPOSE: This clinical trial is studying how well giving cetuximab together with gemcitabine and oxaliplatin works in treating patients with locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the progression-free survival of patients with locally advanced or metastatic pancreatic cancer treated with cetuximab, gemcitabine hydrochloride, and oxaliplatin.

Secondary

* Determine the complete response and partial response in patients treated with this regimen.
* Determine the time to progression in patients treated with this regimen.
* Determine the duration of response in patients treated with this regimen.
* Determine the survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a nonrandomized, open-label, pilot study.

Patients receive cetuximab IV over 1-2 hours on days 1 and 8, gemcitabine hydrochloride IV over 100 minutes on day 1, and oxaliplatin IV over 2-4 hours on day 2. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic cancer
* Locally advanced or metastatic disease
* No active CNS metastases

  * Patients with stable CNS disease, who have undergone radiotherapy within the past 4 weeks and who have been on a stable dose of corticosteroids for > 3 weeks, are eligible

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 mg/dL
* Alkaline phosphatase ≤ 3 times upper limit of normal (ULN) (5 times ULN if known hepatic metastases)
* AST and ALT ≤ 3 times ULN (5 times ULN if known hepatic metastases)
* Creatinine ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 90 days after completion of study treatment
* No significant history of uncontrolled cardiac disease, including any of the following:

  * Uncontrolled hypertension
  * Unstable angina
  * Myocardial infarction within the past 6 months
  * Uncontrolled congestive heart failure
  * Cardiomyopathy with decreased ejection fraction
* No prior severe infusion reaction to a monoclonal antibody
* No active infection or fever ≥ 38.5°C within the past 3 days
* No known hypersensitivity to any components of gemcitabine hydrochloride, oxaliplatin, or to a monoclonal antibody
* No peripheral neuropathy ≥ grade 2
* No known HIV positivity
* No hepatitis B or C infection (active, previously treated, or both)
* No other medical condition, including mental illness or substance abuse, that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy, including surgery
* More than 30 days since prior investigational therapy
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow
* More than 30 days since prior chemotherapy
* No prior chemotherapy for metastatic pancreatic cancer
* Prior fluoropyrimidine as a radiosensitizer allowed
* Prior gemcitabine hydrochloride in the adjuvant setting allowed
* No prior therapy that specifically and directly targets the epidermal growth factor receptor (EGFR) pathway
* No prior allogeneic transplantation
* No other concurrent investigational therapy, chemotherapy, or systemic antineoplastic therapy
* No other concurrent treatment that targets the EGFR
* No other concurrent monoclonal antibody therapy
* No concurrent radiotherapy except for local control of bone pain

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | The cumulative percentage of intent to treat patients who experience disease progression at 1, 2, 3, 4, 5, and 6 months will be characterized with corresponding 95% confidence intervals
  The corresponding progression-free survival curve and cumulative risk of progression as a function of time post treatment initiation will be estimated using the Kaplan-Meier method

SECONDARY OUTCOMES:
Toxicity | Frequency and severity of adverse events according to the NCI CTCAE V 3.0 body system and severity criteria will be described.
Response rate (complete response and partial response) | After every 4th cycle; End of Treatment and Follow-up
  The response rate will be determined by the RECIST criteria. After every 4th cycle; End of Treatment and Follow-up
Duration of response | The time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that recurrence or PD is objectively documented
  the time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that recurrence or PD is objectively documented, taking as reference for PD the smallest measurements recorded since the treatment started
Overall survival | Overall survival will also be estimated using the product-limit method of Kaplan-Meier.
  Overall survival will also be estimated using the product-limit method of Kaplan-Meier.
Time to progression | The time from the start of the treatment until the criteria for disease progression are met
  The time from the start of the treatment until the criteria for disease progression are met, taking as reference the smallest measurements recorded since the treatment started (also referred to in the RECIST criteria as duration of stable disease).

CONTACTS AND LOCATIONS:
Overall Officials: Caio Max S. Rocha Lima, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States